CLINICAL TRIAL: NCT02811653
Title: Motor Slowing and Its Lesion-related Correlates in Alzheimer's Disease
Acronym: TAMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PI2015_843_0003
Record Dates: First submitted 2016-06-16; First posted 2016-06-23 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Alzheimer Disease
Keywords: Motor slowing
MeSH Terms: conditions — Alzheimer Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alzheimer disease (Experimental): Alzheimer disease patients Brain MRI (Magnetic Resonance Imaging) Blood neuropsychological evaluation
  Interventions: Device: Brain MRI; Other: neuropsychological evaluation; Biological: Blood
- control (Active Comparator): Healthy age- and gender-matched volunteers will be recruited into the study from the general population.
  Brain MRI (Magnetic Resonance Imaging) Blood neuropsychological evaluation
  Interventions: Device: Brain MRI; Other: neuropsychological evaluation; Biological: Blood

INTERVENTIONS:
Device: Brain MRI
Other: neuropsychological evaluation
Biological: Blood

SUMMARY:
In AD (Alzheimer disease), the anatomic correlates of attention disorders (as evaluated by motor slowing) have not been thoroughly characterized.

ELIGIBILITY:
Inclusion Criteria:

* Patients

  * Age between 40 and 85
  * French mother tongue
  * Consulting at the Amiens Memory Resource and Research Centre (CMRR) for:
  * MCI, according to Albert et al.'s criteria (Albert et al., 2011)
  * Mild dementia (MMSE>20) due to AD, according to McKhann's criteria (McKhann et al., 2011).
  * Mild dementia due to LBD, according to McKeith et al.'s criteria (McKeith et al., 2005).
  * Mild dementia due to FTLD, according to Rascovsky et al.'s criteria (Rascovsky et al., 2011).
  * Social security coverage
* Healthy controls

  * Healthy age and gender matched volunteers will be recruited into the study from the general population.

Exclusion Criteria:

* Reading or writing difficulties related to a learning disorder or illiteracy.
* A medical history with a potentially significant impact on cognition (non-corrected thyroid disorders or heart failure):

  * NYHA stage IV dyspnoea.
  * respiratory impairment requiring oxygen therapy.
  * liver impairment.
  * kidney failure, progressing neoplastic disease, or past or present alcohol abuse.
* Past or present neurological disorders other than those having prompted consultation in the Memory Clinic:

  * stroke.
  * meningitis or encephalitis.
  * severe head injury.
  * sensorimotor impairments (sensory, proprioceptive, cerebellar and visual impairments).
  * epilepsy (requiring ongoing treatment),
  * psychiatric disorders (other than treated depression).
  * treatment with psychotropic medications (other than anxiolytics or antidepressant withdrawn or initiated in the previous month). Patients with parkinsonian syndrome were examined in the "on-drug" state.
* Impossibility to perform a neuropsychological evaluation or brain MRI.
* Withdrawal from the study at any time, if desired.
* Pregnancy
* Contra-indication to MRI:

  * nerve stimulators
  * cochlear implants
  * ferromagnetic foreign bodies close to nervous structures in the eye or brain
  * cerebral shunts
  * dental appliances
* Legal guardianship or incarceration.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2015-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
median SRT (simple reaction time) to a stimulus (in milliseconds) | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Daniela ANDRIUTA, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France